CLINICAL TRIAL: NCT05136365
Title: The Efficacy and Safety of Xiongdan Wan on Patients With Major Depressive Disorder : a Single-arm, Non-randomized, Open-label Trial
Brief Title: A Study of Xiongdan Wan Treating Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, LI, Huafang, Executive Director of MICT, Shanghai Mental Health Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHXD2021CR2103B
Record Dates: First submitted 2021-11-23; First posted 2021-11-29 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Xiongdan Wan is used in patients diagnosed with Major Depressive Disorder.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Xiongdan Wan group (Experimental): Xiongdan Wan is used in patients diagnosed with Major Depressive Disorder. The daily dose (1350mg per day) should be strictly controlled according to the experimental design.
  Interventions: Drug: Xiongdan Wan

INTERVENTIONS:
Drug: Xiongdan Wan — Xiongdan Wan is used as 450mg three times a day after meals with water for 8 weeks. The daily dose (e.g. 450mg/bag, 3 times/day) should be strictly controlled according to the experimental design. Patients should take medicine regularly every day under the guidance of doctors.

SUMMARY:
This is a prospective, single-arm, open-label study to evaluate the safety and efficacy of Xiongdan Wan monotherapy in patients with Major Depressive Disorder(MDD), conducted in Shang Hai Mental Health Center. Following a screening period, subjects who meet the entry criteria will be treated with 450mg Xiongdan Wan pills three times daily for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the Diagnostic and Statistical Manual of Mental Disorder, Fourth Edition Text Revision (DSM-IV-TR) criteria for Major Depressive Disorder (MDD): a single or recurrent episode without psychotic features. Codes are as follows: F32.0, F32.1, F32.2, F33.0, F33.1, F33.2.
2. Outpatients.
3. Male or female subjects aged 18-65 years.
4. HAMD-17 score of the baseline period and screening period is 18-24.
5. Women of childbearing potential must be willing to use acceptable methods of contraception throughout the study period and the following one month.
6. The patient fully understands and signs the informed consent form.

Exclusion Criteria:

1. Patient has survived a suicide attempt or has acute suicidal tendencies (HAMD-17 Item3 ≥3).
2. Comorbidity according to DSM-IV-TR, axis-I except for major depressive disorder.
3. HAMD-17 reduction ratio ≥25% within one week from the screening to the baseline period.
4. Depressive episode secondary to psychiatric illness or somatic disease.
5. Serious and unstable diseases such as cerebrovascular disease; liver and kidney disease; disease of internal secretion (abnormal thyroid function); hemopathy; seizures, or other encephalopathies.
6. History of alcohol or drug abuse over the last 6 months.
7. Allergic history to Xiongdan Wan, or serious drug allergic history.
8. Pregnant or lactating women and women of childbearing potential throughout the study period; men who have the desire of fertility within six months.
9. Clinically significant changes in ECG or laboratory tests, including >1.5 times the upper limit of normal liver function; over the limit of normal renal function and blood sugar; abnormal cardiac troponins; obvious abnormity in the thyroid function.
10. Treatment with modified electroconvulsive therapy (MECT) or repetitive transcranial magnetic stimulation (rTMS) in the past three months.
11. Treatment with a systematic psychological treatment in the past three months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change in the Montgomery-Asberg Depression Rating Scale (MADRS) score compared with baseline at the end of study. | 8 weeks
  The main objective is to explore whether Xiongdan Wan improve the MDD symptoms after 8 weeks of treatment, and investigators assess the scale at week 1, 2, 4, 8.

SECONDARY OUTCOMES:
Effective treatment | 8 weeks
  Montgomery-Asberg Depression Rating Scale (MADRS) or Hamilton Depression Rating Scale （HAMD-17）reduction ratio ≥50% reductive ratio [（Baseline score- Endpoint score）／Baseline score]×100%
Clinical remission rate | 8 weeks
  Patients in remission at the end of the study will be summarized, Montgomery-Asberg Depression Rating Scale (MADRS) score ≤12 or Hamilton Depression Rating Scale （HAMD-17）≤7.
The Montgomery-Asberg Depression Rating Scale (MADRS) reduction ratio | 8 weeks
  MADRS reduction ratio is used to evaluate the effectiveness of the treatment and investigators assess the scale at week 1, 2, 4, 8.
The Hamilton Depression Rating Scale (HAMD-17) reduction ratio | 8 weeks
  HAMD-17 reduction ratio is used to evaluate the effectiveness of the treatment and investigators assess the scale at week 1, 2, 4, 8.
Change in the total score of the Hamilton Anxiety Scale(HAMA) | 8 weeks
  The change of HAMA is used to evaluate the effectiveness of the treatment and investigators assess the scale at week 1, 2, 4, 8.
Change in total score of the Clinical Global Impression scale(CGI) | 8 weeks
  The change of CGI is used to evaluate the effectiveness of the treatment and investigators assess the scale at week 1, 2, 4, 8.

CONTACTS AND LOCATIONS:
Overall Officials: Huafang LI, MD, PHD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No